CLINICAL TRIAL: NCT03648112
Title: Intervention Study - Physiological Short-term and Long-term Effects of Regularly Consumption of Beta-glucan From Barley and Oats on the Glucose and Lipid Metabolism and Satiety
Brief Title: Effects of Beta-glucan From Barley and Oats on Glucose and Lipid Metabolism, and Satiety
Acronym: gLUCAn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, Leader of the Junior Research Group Nutritional Concepts, University of Jena
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H7_18
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Lipid Metabolism; Glucose Metabolism; Satiety
Keywords: dietary fibres; ß-glucan; low-density-lipoprotein-cholesterol; insulin; fasting glucose; microbiota
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intervention 1 (Active Comparator): Intervention 1: Crude oat flakes (dietary supplement) 80 g of crude oat flakes contain 4 g ß-glucan. According to the current Health Claim, 4 g ß glucan are necessary to achieve a reduction of the postprandial glycemic answer and a reduction of the cholesterol concentration in hypercholesterolinaemic patients.
  The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of crude oat flakes.
  Interventions: Dietary Supplement: Intervention 1
- Intervention 2 (Active Comparator): Roasted oat flakes (dietary supplement) 80 g of roasted oat flakes contain 4 g ß-glucan. According to the current Health Claim, 4 g ß-glucan are necessary to achieve a reduction of the postprandial glycemic answer and a reduction of the cholesterol concentration in hypercholesterolinaemic patients.
  These oat flakes were roasted at 150°C for 20 minutes.
  The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of roasted oat flakes.
  Interventions: Dietary Supplement: Intervention 2
- Intervention 3 (Active Comparator): Crude barley flakes (dietary supplement) 80 g of crude oat flakes contain 4 g ß-glucan. According to the current Health Claim, 4 g ß-glucan are necessary to achieve a reduction of the postprandial glycemic answer and a reduction of the cholesterol concentration in hypercholesterolinaemic patients.
  The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of crude barley flakes
  Interventions: Dietary Supplement: Intervention 3
- Intervention 4 (Active Comparator): Roasted barley flakes (dietary supplement) 80 g of roasted oat flakes contain 4 g ß-glucan. According to the current Health Claim, 4 g ß-glucan are necessary to achieve a reduction of the postprandial glycemic answer and a reduction of the cholesterol concentration in hypercholesterolinaemic patients.
  The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of roasted barley flakes.
  Interventions: Dietary Supplement: Intervention 4
- control (Placebo Comparator): White toastbread (control) (dietary supplement) White toastbread was chosen because of its low fibre content. To achieve the same energy value (kcal) as 80 g cereal flakes the participants have to consume four slices of white toastbread.
  The study participants receive recipes for breakfast for 21 days. The recipes imply four slices of white toastbread.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Intervention 1 — The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of crude oat flakes per day.
  Other Names: Crude oat flakes
  Arms: Intervention 1
Dietary Supplement: Intervention 2 — The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of roasted oat flakes per day.
  Other Names: Roasted oat flakes
  Arms: Intervention 2
Dietary Supplement: Intervention 3 — The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of crude barley flakes per day.
  Other Names: Crude barley flakes
  Arms: Intervention 3
Dietary Supplement: Intervention 4 — The study participants receive recipes for breakfast for 21 days. The recipes imply 80 g of roasted barley flakes per day.
  Other Names: Roasted barley flakes
  Arms: Intervention 4
Dietary Supplement: Control — White toastbread (control) (dietary supplement) White toastbread was chosen because of its low fibre content. To achieve the same energy value (kcal) as 80 g cereal flakes the participants have to consume four slices of white toastbread.
  The study participants receive recipes for breakfast for 21 days. The recipes imply four slices of white toastbread.
  Other Names: White toast bread
  Arms: control

SUMMARY:
The interventional study will evaluate the effects of a regularly consumption of barley and oat flakes in crude and roasted form on the glucose and lipid metabolism as well as the postprandial saturation. Moreover, the study will evaluate the effect of a regularly consumption of barley and oat flakes on the glucose and lipid metabolism over a period of three weeks.

All participants will run through each intervention (cross-over design). Inbetween these intervention periods there will be wash-out phases. In total there will be four interventions: crude oat flakes, roasted oat flakes, crude barley flakes and roasted barley flakes. The comparison will be made against white toastbread. The study participants will visit the study centrum before and after each intervention over an entire period of 27 weeks.

DETAILED DESCRIPTION:
The interventional study will evaluate the effects of a regularly consumption of barley and oat flakes in crude and roasted form on the glucose and lipid metabolism as well as the postprandial saturation. Moreover, the study will evaluate the effect of a regularly consumption of barley and oat flakes on the glucose and lipid metabolism over a period of three weeks.

By applying the cross-over design, all participants will run through each intervention. In total there will be four interventions: crude oat flakes, roasted oat flakes, crude barley flakes and roasted barley flakes. Each intervention period will last three weeks and will be separated by wash-out phases which also will last three weeks. The comparison will be made against white toastbread, which will be the fifth intervention. The entire duration of the study will be 27 weeks (5x 3 weeks intervention + 4x 3 weeks wash-out phases inbetween).

The participants will visit the study centrum before and after each intervention for examinations and for taking blood samples. During the examination the participants will receive a test-meal to evaluate postprandial blood glucose and insulin levels. Moreover, the kinetic of hormones that influence the satiety will be evaluated. In addition to the examination of blood samples, the microbiota of feces will be examined.

During the intervention periods the participants will receive recipes for breakfast for 21 days. In these recipes 80 gram oat or barley flakes or four slices of white toastbread will be included.

The study will provide data about the association between different processed cereals and measurable markers reflecting glucose and lipid metabolism as well as their influence on hormones of satiety and microbiota.

ELIGIBILITY:
Inclusion Criteria:

* LDL-cholesterol ≥ 120 mg/dl (≥ 3 mmol/l)
* Typical western diet

Exclusion Criteria:

* intake of lipid-lowering medications
* gastrointestinal diseases
* diabetes mellitus type I and II
* familial hypercholesterolemia
* intake of additional dietary supplements (especially ß-glucan capsules, high-fibre compounds)
* pregnancy, lactation
* appreciable food allergies/intolerances
* patient´s request or if patient compliance with the study protocol is doubtful

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No] [mmol/L]
  LDL cholesterol [mmol/L]

SECONDARY OUTCOMES:
total cholesterol | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No] total cholesterol, LDL cholesterol, HDL cholesterol, triacylglycerides (TAG) [mmol/L]
  total cholesterol [mmol/L]
HDL cholesterol | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No] total cholesterol, LDL cholesterol, HDL cholesterol, triacylglycerides (TAG) [mmol/L]
  HDL cholesterol [mmol/L]
triacylglycerides | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No] total cholesterol, LDL cholesterol, HDL cholesterol, triacylglycerides (TAG) [mmol/L]
  triacylglycerides [mmol/L]
HOMA-index | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  HOMA-index
fasting blood glucose | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  fasting blood glucose [mg/dl]
kinetic of glycemic answer | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  blood glucose (mg/dl; timepoints: 0, 30, 60, 120 and 180 min) after a test meal)
kinetic of satiety hormones | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  Ghrelin, GLP1, peptide YY (timepoints: 0, 30, 60, 120 and 180 min) after a test meal)
short chain fatty acids in fecal water | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  short chain fatty acids (SCFA; %) , pH value, composition of microbiome
composition of microbiome | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  composition of microbiome [%]
blood pressure | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  systolic and diastolic blood pressure [mmHg]
height | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  Height [m]
weight | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  Weight [kg]
body-mass index | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  body-mass index [kg/m2]
bioelectrical impedance analysis | [Time Frame: change from baseline to 3 weeks intervention] [Safety Issue: No]
  bioelectrical impedance analysis (%)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dawczynski, PhD, Principal Investigator — University of Jena; Stefan Lorkowski, PhD, Principal Investigator — University of Jena
Locations (1):
- Friedrich-Schiller-University, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reiners S, Hebestreit S, Wedekind L, Kiehntopf M, Klink A, Rummler S, Glei M, Lorkowski S, Schlormann W, Dawczynski C. Effect of a regular consumption of traditional and roasted oat and barley flakes on blood lipids and glucose metabolism-A randomized crossover trial. Front Nutr. 2023 Feb 2;10:1095245. doi: 10.3389/fnut.2023.1095245. eCollection 2023. PMID 36819683
- See also: Study results — https://www.frontiersin.org/articles/10.3389/fnut.2023.1095245/full